CLINICAL TRIAL: NCT00503022
Title: A Randomized, Double-Masked, Multi-Center Phase I Study of 6 Months Duration to Assess the Safety and Tolerability of Intravenous ACZ885 in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: Safety and Tolerability of an Intravenous Infusion of ACZ885 in Patients With Wet Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885F2201
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Wet Age-Related Macular Degeneration
Keywords: Wet age-related macular degeneration; ACZ885
MeSH Terms: interventions — canakinumab

INTERVENTIONS:
Drug: ACZ885

SUMMARY:
This study evaluates the tolerability and safety of a single intravenous infusion of ACZ885. It also explores the efficacy of the compound in central macular edema and visual acuity in patients with wet age-related macular edema.

ELIGIBILITY:
Inclusion criteria:

* Male or female ≥ 50 years old, with aged related macular degeneration
* Patients with subfoveal choroidal neovascularization secondary to age-related macular degeneration

Exclusion criteria:

* Active intraocular inflammation or ocular infection in the study eye
* Eye disease that may result in visual loss during the study
* Chronic therapy with topical, local or systemic corticosteroids.
* Pregnant or nursing (lactating) women.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-07

PRIMARY OUTCOMES:
Rates of adverse events and serious adverse events, as well as changes in ophthalmic evaluations, laboratory values, electrocardiograms (ECGs) and vital signs over 6 months, following single intravenous infusion of ACZ885.

SECONDARY OUTCOMES:
Changes in central macular edema from Baseline up to Month 6 Changes in best-corrected visual acuity from Baseline up to Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Novartis EH 001 862 778 8300, Study Chair — COREC,UK
Locations (8):
- Bern, Switzerland
- United Kingdom (7):
  - Belfast, Northern Ireland
  - Bristol
  - Liverpool
  - London
  - Nottingham
  - Southampton
  - Wolverhampton